CLINICAL TRIAL: NCT05784480
Title: Relevance of Reversible Causes During OHCA (Rebecca Study)
Acronym: REBECCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Seibersdorf Labor GmbH (Industry); Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Responsible Party: Principal Investigator, Christina Hafner, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rebecca Vienna
Record Dates: First submitted 2023-01-06; First posted 2023-03-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Cardiopulmonary Arrest
Keywords: Intoxication; Prehospital POCUS; CPR; Sonography; Blood gas analysis; Cardiac arrest; OHCA; Reversible causes; Tele-support; Checklist; Prehospital emergency physician; Emergency medicine
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation of reversible causes using digital checklist and diagnostic support (Other)
  Interventions: Diagnostic Test: Checklist for evaluation of reversible causes

INTERVENTIONS:
Diagnostic Test: Checklist for evaluation of reversible causes — Prehospital evaluation by checklist and diagnostic testing for reversible causes of OHCA using point-of-care blood gas analysis, saliva toxicological screen and ultrasound and post-hoc toxicological analysis of blood using mass spectrometry
  Other Names: Venipuncture for toxicological screening; Point-of-Care blood gas analysis; Point-of-Care saliva toxicological screen; Point-of-care ultrasound

SUMMARY:
Management of the reversible causes in cardiac arrest is fundamental for successful treatment of out-of-hospital cardiac arrests. Point-of-care diagnostics as prehospital emergency ultrasound, blood gas analysis and toxicological screening support the diagnostic process of evaluating potential reversible causes. Digital tools provide support of a structured approach. This study aims to evaluate the frequency of reversible causes during OHCA as well as specific interventions due to these findings. Furthermore, CPR performance (hands-off, ROSC, 30-day mortality) and cognitive load of the prehospital emergency physician will be investigated. In total 100 patients with OHCA will be included in this study. Identification of reversible causes will be performed upon a structured protocol using an interactive checklist. Cognitive load of emergency physician as well as CPR parameter (frequency of reversible causes, hands-off, ROSC, 30-day mortality) will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prehospital cardiac arrest, where POCUS, blood gas analysis as well as screening for intoxication can integrated in ALS rhythm without delay of life-saving treatment or transportation will be included.

Exclusion Criteria:

* Patients will be excluded under the age of 18, or if POCUS, blood gas analysis will lead to a delay of live-saving treatment or transportation. Furthermore, pregnant patients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of reversible causes in OHCA and alterations of treatment | up to 30 days
  The primary outcome of this study evaluates the frequency of reversible causes during OHCA.

SECONDARY OUTCOMES:
Frequency of ROSC | up to 30 days
  Any prehospital ROSC/sustained ROSC/in-hospital ROSC
30-day mortality | up to 30 days
  rate of mortality within 30 days in case of hospital admission
Hands-off time | During study completion, up to 120 min
  Hands-off time during process of identification of reversible causes
Cognitive load | 1 year (evaluation in documentation phase after CPR)
  NASA Task Load Index evaluated by the prehospital emergency physician after rescue mission

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Anesthesiology and Intensive Care Medicine Department - Medical University of Vienna, Vienna, Austria
  - Department of Anesthesia, General Intensive Care and Pain Management,Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No